CLINICAL TRIAL: NCT04940286
Title: Phase II Study of Neoadjuvant Gemcitabine, Nab-paclitaxel, Durvalumab (MEDI4736) (Anti-PD-L1), and Oleclumab (Anti-CD73) in the Treatment of Resectable/Borderline Resectable Primary Pancreatic Adenocarcinoma
Brief Title: Gemcitabine, Nab-paclitaxel, Durvalumab, and Oleclumab Before Surgery for the Treatment of in Resectable/Borderline Resectable Primary Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0898; NCI-2021-05721 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0898 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma; Resectable Pancreatic Adenocarcinoma; Stage IA Pancreatic Cancer AJCC v8; Stage IB Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (durvalumab, oleclumab, nab-paclitaxel, gemcitabine) (Experimental): Patients receive durvalumab IV over 1 hour on day 1, oleclumab IV over 1 hour, nab-paclitaxel IV, and gemcitabine IV over 1 hour over 30-40 minutes on days 1 and 15. Treatment repeats every 28 days for 2-6 cycles. Within 4-8 weeks after completion of last cycle of treatment, patients undergo surgical resection. After surgical resection, patient may receive adjuvant therapy with durvalumab and oleclumab, durvalumab, oleclumab, gemcitabine, and nab-paclitaxel, other chemotherapy, or observation only at the discretion of the treating physician.
  Interventions: Biological: Durvalumab; Drug: Gemcitabine; Drug: Nab-paclitaxel; Biological: Oleclumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
Biological: Oleclumab — Given IV
  Other Names: Anti-CD73 Monoclonal Antibody MEDI9447; MEDI9447

SUMMARY:
This phase II trial studies the effects of gemcitabine, nab-paclitaxel, durvalumab, and oleclumab in treating patients with primary pancreatic cancer that may be able to be removed by surgery (resectable/borderline resectable). Chemotherapy drugs, such as gemcitabine and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as durvalumab and oleclumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving gemcitabine, nab-paclitaxel, durvalumab, and oleclumab may help control the disease in patients with resectable/borderline resectable primary pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimation of major pathological response (MPR) rate (=< 5% viable tumor cells).

II. Assess the safety of combining immunotherapy (durvalumab and oleclumab) with gemcitabine/nab-paclitaxel as neoadjuvant therapy.

EXPLORATORY OBJECTIVES:

I. Explore the changes in various immune parameters, including PD-L1 and PD-1 expression in the tumor, during treatment and correlate with efficacy outcomes with the goal of biomarker discovery.

II. Radiographic response rate and CA19-9 response to neoadjuvant therapy. III. Estimate the relapse-free survival (RFS) and overall survival (OS) in enrolled subjects who undergo surgical resection.

IV. Estimate the frequency of intraoperative and postoperative complications in these patients treated with neoadjuvant therapy.

V. Impact of adjuvant durvalumab/oleclumab +/- gemcitabine/nab-paclitaxel on circulating tumor-derived deoxyribonucleic acid (ctDNA) kinetics.

OUTLINE:

Patients receive durvalumab intravenously (IV) over 1 hour on day 1, oleclumab IV over 1 hour, nab-paclitaxel IV, and gemcitabine IV over 1 hour over 30-40 minutes on days 1 and 15. Treatment repeats every 28 days for 2-6 cycles. Within 4-8 weeks after completion of last cycle of treatment, patients undergo surgical resection. After surgical resection, patient may receive adjuvant therapy with durvalumab and oleclumab, durvalumab, oleclumab, gemcitabine, and nab-paclitaxel, other chemotherapy, or observation only at the discretion of the treating physician.

After completion of study treatment, patients are followed up 28 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent includes any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Age >= 18 years at time of study entry
* Has histologically or cytologically confirmed resectable or borderline resectable pancreatic adenocarcinoma per MD Anderson criteria (borderline patients based upon reconstructable superior mesenteric vein/portal vein [SMV/PV] involvement or reconstructable hepatic artery involvement are allowed)
* Has received no prior anti-cancer therapy for pancreatic adenocarcinoma
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count 1.5 x (>= 1500 per mm^3)
* Platelet count >=100 x 10^9/L (>= 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician. Subjects requiring biliary decompression, biliary stent, or drainage using percutaneous trans-hepatic cholangiogram are allowed (patients with a declining bilirubin status post stent placement are eligible with serum bilirubin =< 2.5 x institutional ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN
* Measured creatinine clearance (CL) > 40 mL/min or calculated creatinine CL> 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Has evidence of post-menopausal status or negative urinary- or serum pregnancy test for female, pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or if they underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up
* Must have a predicted life expectancy of at least 6 months
* Is willing to undergo mandatory research esophagogastroduodenoscopy/endoscopic ultrasound for fine-needle aspiration (exceptions to this eligibility can be discussed with principal investigator [PI] and will be considered on a case-by-case basis)
* Has body weight of > 35 kg

Exclusion Criteria:

* Participated in another clinical study with an investigational product during the last 4 weeks from the first dose of this study's treatment
* May need preoperative radiation therapy (as determined per the treating medical team: medical oncologist and/or surgical oncologist at time of study enrollment)
* Is concurrently enrolled in another clinical study (patient is eligible if the study is an observational (non interventional) study or if enrollment is during the follow-up period of an interventional study
* Has definitive evidence of metastatic disease per radiographic assessment
* Is receiving any concurrent chemotherapy, investigational product (IP), or biologic- or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* Had a major surgical procedure within 28 days prior to the first dose of IP (PORT placement does not count; if classification is uncertain, discuss with PI)
* Has history of allogenic organ transplantation
* Has an active or previously documented autoimmune or inflammatory disorder (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [diverticulosis is not an excluding factor], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion (and do not exclude patients from participation):

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Patients having any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years (allowed only after consultation with the study physician)
  * Patients with celiac disease controlled by diet alone
* Has uncontrolled intercurrent illness, including but not limited to, ongoing or active infection; symptomatic congestive heart failure; uncontrolled hypertension; unstable angina pectoris; cardiac arrhythmia; interstitial lung disease; serious chronic gastrointestinal conditions associated with diarrhea; or psychiatric illness/social situations that would limit compliance with study requirements, would substantially increase risk of incurring adverse events (AEs), or would compromise the ability of the patient to give written informed consent
* Has a history of another primary malignancy. Patients having the following are still eligible:

  * Malignancy treated with curative intent, no known active disease >= 5 years before the first dose of IP, and low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Has a history of leptomeningeal carcinomatosis
* Has a history of active primary immunodeficiency
* Has active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), or hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (hepatitis C virus [HCV]) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Is currently using or previously used immunosuppressive medication within 14 days before the first dose of durvalumab. The following medications are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Has received live attenuated vaccine within 30 days prior to the first dose of IP. Note: patients, if enrolled, should not receive live vaccine while receiving IP or during the 30 days after the last dose of IP
* Is a female and pregnant or breastfeeding; or is a male or female of reproductive potential who is not willing to employ effective birth control from time of screening to 90 days after the last dose of durvalumab and oleclumab monotherapy
* Has a known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Previously received clinical-trial treatment with durvalumab or oleclumab regardless of treatment arm assignment
* Has laboratory evidence of hypercalcemia (>= 11 mg/dL [in presence of normal albumin]) and/or hyperphosphatemia (>= 5.5 mg/dL)
* Has a history of venous thrombosis within the past 3 months prior to scheduled first dose of study treatment and is not receiving fully dosed anticoagulation; or has symptomatic venous thrombosis and symptoms have not improved
* Has a prior history of myocardial infarction, transient ischemic attack, or stroke within the past 3 months prior to the scheduled first dose of study treatment
* Is unsuitable to participate in the study or is unlikely to comply with study procedures, restrictions and requirements (per judgment by the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate (=< 5% viable tumor cells) | Up to 2 years
  A Chi square- or Fisher's exact test will be used to evaluate the association between patient prognostic factor and response. Paired t-tests will be used to determine parameter changes before and after surgery in various immune-based conditions.
Incidence of adverse events | Up to 2 years
  Assessed using the Common Terminology Criteria for Adverse Events Version 5.0.

OTHER OUTCOMES:
Radiographic response rate | Up to 2 years
Recurrence-free survival | Up to 2 years
  Will be estimated using the method of Kaplan and Meier and the log-rank test.
Overall survival | Up to 2 years
  Will be estimated using the method of Kaplan and Meier and the log-rank test.
Frequency of intraoperative and postoperative complications | Up to 2 years
Change in circulating tumor deoxyribonucleic acid (ctDNA) levels | Baseline to 2 years
  Patient ctDNA levels may be tracked at various time-points during the study to identify patterns of change following therapy with durvalumab and oleclumab and its association to treatment benefit in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon G Smaglo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT04940286/ICF_000.pdf